CLINICAL TRIAL: NCT06732492
Title: RD13-02 Cell Injection in Patients with Relapsed or Refractory CD7-Positive Natural Killer/T Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-RD13-02-01
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: NK T-Cell Lymphoma; CART Therapy; CD7-positive Relapsed/Refractory Lymphoid Hematologic Malignancies
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RD13-02 cell infusion (Experimental): RD13-02 cells targeting CD7 were injected intravenously
  Interventions: Drug: RD13-02 cell infusion

INTERVENTIONS:
Drug: RD13-02 cell infusion — CAR-T cells
  Other Names: universal CD7 CAR-T cells

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD7 Chimeric Antigen Receptor-T(CAR-T) therapy for patients with CD7-positive relapsed or refractory natural killer/T cell lymphoma, and to evaluate the pharmacokinetics of CD7 CAR-T in patients。

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-70
2. Diagnosis of r/r NK/T lymphoma.
3. CD7 positive expression
4. Bone marrow lymphoblasts ≥5% by morphologic evaluation at screening
5. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min, Serum alanine aminotransferase(ALT)/aspartate aminotransferase(AST) < 3×upper limit of normal, Total bilirubin < 1.5×upper limit of normal or ≤1.5mg/dl
6. Left ventricular ejection fraction ≥ 50% .
7. Baseline oxygen saturation ≥ 92% on room air.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
9. The estimated survival time is more than 3 months.
10. Subjects or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Subjects with concomitant genetic syndromes associated with bone marrow failure states.
2. Isolated extramedullary lesions
3. Subjects with some cardiac conditions will be excluded.
4. With uncontrolled active central nervous system leukemia (CNSL), cerebrospinal fluid grade Central Nervous System3(CNS3).
5. History of traumatic brain injury, consciousness disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic disease, which might compromise the ability of the subject to compliance with the obligations under the protocol.
6. History of malignancy other than non-melanoma skin cancer or carcinoma.
7. Primary immune deficiency.
8. Presence of uncontrolled infections.
9. Subjects with some anticancer therapy before CAR-T infusion will be excluded.
10. Active uncontrolled acute infections.
11. Known history of infection with human immunodeficiency virus (HIV); active or latent hepatitis B, hepatitis C and syphilis.
12. Subjects who are receiving systemic steroid therapy prior to screening.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Evaluate at 4 weeks after CAR-T infusion
  The proportion of patients with complete response (CR) /complete response with incomplete blood cell recovery (CRi)

SECONDARY OUTCOMES:
Duration of remission (DOR) | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Event-free survival (EFS) | Up to 1 years after CAR-T infusion
  The time from first achieving CR/CRi to relapse or death
Overall survival (OS) | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No